CLINICAL TRIAL: NCT03499522
Title: Situation and Characteristics of Pain in Patients With Congenital Coagulopathies in Spain
Brief Title: Pain in Patients With Congenital Coagulopathies
Acronym: He-PainSit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Real Fundación Victoria Eugenia
Other Study IDs: He-Pain Situation
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Hemophilia Arthropathy
Keywords: Hemophilic arthropathy; Pain; Functional Disease Present; Quality of life; Anxiety; Stress; Coping strategies
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: 80 patients with congenital coagulopathies (hemophilia A and B, and von Willebrand's disease), of legal age, will be included in the study. Patients will be recruited in six centers, from different regions of Spain.
  The inclusion criteria to participate in the present study are patients: with a medical diagnosis of congenital coagulopathies (hemophilia A and B, or von Willebrand's disease); adults; in a prophylactic or on demand regimen with FVIII / FIX concentrates; and that they have signed the informed consent document.
  On the other hand, those patients with: neurological or cognitive alterations that impede the comprehension of the questionnaires will be excluded from the study; inability to walk autonomously or with an orthosis; and without access to digital media to complement the measuring instruments.
  Interventions: Other: Observational group

INTERVENTIONS:
Other: Observational group — The dependent variables (pain, quality of life, anxiety and coping strategies) and the outcome measures used to measure these variables will be:
  * Numerical scale of pain
  * Short Form 36 Health Survey [SF-36].
  * State-Trait Anxiety Inventory [STAI].
  * Tampa Scale of Kinesiophofia [TSK-11SV].
  * Pain catastrophizing scale [PCS].
  * Coping Strategies Questionnaire [CSQ].

SUMMARY:
Introduction. The development of joint hemorrhages in patients with congenital coagulopathies favor the development of an intra-articular, degenerative and progressive lesion (hemophilic arthropathy). Pain is one of the main clinical manifestations of hemophilic arthropathy and is related to the development of disability and a worse quality of life.

Objective. Observe the characteristics of pain, coping models and the perception of quality of life in patients with congenital coagulopathies.

Study design. Observational, cross-sectional and multi-center study. Method. 80 patients with congenital coagulopathies (hemophilia A and B, and von Willebrand's disease), of legal age, will be included in the study. Patients will be recruited in six centers, from different regions of Spain. The study variables and measurement instruments used will be: pain perception (numerical pain scale, Tampa Scale of kinesiophobia and Pain Catastrophizing Scale); perception of quality of life (Short Form -36 questionnaires); anxiety (State-Trait Anxiety Questionnaire); coping strategies (Coping Strategy Questionnaire); and disease perception (Illness behaviour questionnaire and Revised Illness Perception Questionnaire). A descriptive statistical analysis of the dependent and independent variables will be carried out. In the same way, the correlations between the variables and the characteristics of the subjects will be analyzed according to age, the type of coagulopathy and the degree of sequelae.

Expected results. Observe the characteristics of pain, its coping models and its implication in the quality of life in patients with congenital coagulopathies, and evaluate the independent variables related to the perception of pain.

DETAILED DESCRIPTION:
Objectives:

Main objective: to observe the characteristics of pain, its coping models and its implication in the quality of life in patients with congenital coagulopathies. Secondary objectives: to evaluate the degree of kinesiofobia and catastrophism in patients with congenital coagulopathies; analyze the perception of quality of life, of disease and of anxiety in patients with hemophilia and von Willebrand's disease of age; and to identify the ingestion and administration of analgesic drugs in patients with hemophilia or von Willebrand's disease for the control of pain.

Design of the investigation Describe the type of study, methodology, research variables Cross-sectional and multicentric observational study, carried out in patients with congenital coagulopathies, with the aim of knowing the characteristics of pain, its coping strategies and its implications for quality of life.

Collection of information Instruments and data collection process

* Numerical scale of pain. The patient assigns pain a numerical value between 0 and 10. With this scale pain is considered a simple one-dimensional concept and is measured only according to its intensity. The scale is discrete, not continuous.
* Short Form 36 Health Survey (SF-36). Health questionnaire that measures the quality of life related to health. Generic instrument consisting of 36 questions, covering 8 dimensions (physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role and mental health of the patient).
* State-Trait Anxiety Inventory (STAI). Generic instrument that assesses the current level of anxiety and the predisposition of the person to respond to stress. It consists of two sections that let you know how you feel at a certain time and how you feel in general. The score for each scale can range from 0-30, indicating higher scores, higher levels of anxiety.
* Tampa Scale of kinesiophobia (TSK-11SV). Through this scale the fear of movement of the patients included in the study will be evaluated. This self-report measure contains 17 items on fear of movement and recurrence of a new lesion. Four of the items have a negative wording and carry an inverse notation. The scores of the different items evaluated are added to give a total score, where the highest values reflect a greater fear of injury or relapse of the same.
* Pain catastrophizing scale (PCS). Self-administered scale of 13 items used to assess the 3-dimensional pain-mapping construct: rumination, magnification and hopelessness. Low scores indicate a low catastrophization, and high values, high catastrophization.
* Coping Strategies Questionnaire (CSQ). Questionnaire composed of 42 items grouped in 7 scales of 6 items each. Each item is scored according to a scale of 7 points: deviation of attention, reinterpretation of pain sensations, ignorance of pain sensations, self-assertive coping, prayer and hope, catastrophism and increased level of activity.

Subjects of the study Number and characteristics of the sample. The inclusion criteria to participate in the present study are patients: with a medical diagnosis of congenital coagulopathies (hemophilia A and B, or von Willebrand's disease); adults; in a prophylactic or on demand regimen with FVIII / FIX concentrates; and that they have signed the informed consent document. On the other hand, those patients with: neurological or cognitive alterations that impede the comprehension of the questionnaires will be excluded from the study; inability to walk autonomously or with an orthosis; and without access to digital media to complement the measuring instruments.

It is expected to recruit a total of 80 patients for inclusion in the study. The sample size is justified with respect to the prevalence of patients with hemophilia (2039 patients with hemophilia A and B in Spain). Based on the established selection criteria (n = 678, according to the census of the Spanish Federation of Hemophilia) the sample size at the national level would be 151, with a level of confidence or 95% confidence and an expected proportion of dropouts from the fifteen%. Thus, for the 6 regions of Spain where the study will be developed, a sample of 80 patients is established for the established study period (April to December 2018).

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical diagnosis of congenital coagulopathies: hemophilia A, hemophilia B, or von Willebrand's disease
* Patients over 18 years of age
* Patients in a prophylactic or on demand regimen with FVIII / FIX concentrates
* Patients that have accepted the informed consent document.

Exclusion Criteria:

* Patients with neurological or cognitive disorders that prevent the comprehension of the questionnaires
* Patients without capacity to walk autonomously or with orthosis
* Patients without access to digital media to complement the measuring instruments.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia attending in six hemophilia Associations into Spanish Federation of Hemophilia (Fedhemo).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Perception of joint pain | Screening visit
  Measurement with numerical scale of pain. The patient must assign pain to a numerical value between two extreme points (0 to 10). Although the subject is asked to use numerical values to indicate the level of pain, the use of keywords, as well as previous instructions, are necessary if the investigators expect the patient to conceptualize their pain in numerical terms. The scale is discrete, not continuous, but to perform statistical analyzes, equal intervals can be assumed between categories.

SECONDARY OUTCOMES:
Perception of pain coping strategies | Screening visit
  Measurement with Coping Strategies Questionnaire [CSQ]. Questionnaire composed of 42 items grouped in 7 scales of 6 items each, plus 2 items referring to the control exercised over pain and the ability to reduce it. Each item is scored according to a scale of 7 points (0 = never, 3 = sometimes, 6 = always). The scales included in this measuring instrument are: deviation of attention, reinterpretation of pain sensations, ignoring pain sensations, self-assertive coping, prayer and hope, catastrophism and increased level of activity.
Perception of quality of life | Screening visit
  Measurement with Short Form 36 Health Survey [SF-36]. This health questionnaire is one of the most widely used, validated and translated instruments in the field of measuring the quality of life related to health. The SF-36 health questionnaire is a generic instrument consisting of 36 questions, which provides a profile of the health status and is applicable to both patients and the healthy population. The questionnaire covers 8 dimensions: physical functioning, physical role, corporal pain, general health, vitality, social functioning, emotional role and mental health of the patient.
Perception of anxiety | Screening visit
  Measurement with State-Trait Anxiety Inventory [STAI]. This generic measurement instrument evaluates the current level of anxiety and the predisposition of the person to respond to stress. The STAI scale consists of two sections: the A-state scale contains 20 elements with which the patient can express how they feel at a given time and in the A-trait sscala, which also includes 20 elements, the subject can indicate how they feel. feel in general. The score for each scale can range from 0-30, indicating higher scores, higher levels of anxiety.
kinesiophobia | Screening visit
  Measurement with Tampa Scale of kinesiophobia [TSK-11SV]. Through this scale the fear of movement of the patients included in the study will be evaluated. This self-report measure contains 17 items on fear of movement and recurrence of a new lesion. Four of the items have a negative wording and carry an inverse notation. The scores of the different items evaluated are added to give a total score, where the highest values reflect a greater fear of injury or relapse of the same.
Perception of pain catastrophizing | Screening visit
  Measurement with Pain catastrophizing scale [PCS]. This self-administered scale of 13 items is one of the most used to assess the construct catrastofización before pain. It includes 3 dimensions: rumination, magnification and despair. The theoretical range of the instrument is between 13 and 62, indicating low scores a low catastrophization, and high values, high catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta Barriuso, Principal Investigator — Royal Victoria Eugenia Foundation

IPD SHARING:
Plan to Share IPD: No